CLINICAL TRIAL: NCT05024721
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Phase Ⅲ Study to Evaluate the Efficacy and Safety of HIP2101 in Patients With Acute or Chronic Gastritis
Brief Title: Study to Evaluate the Efficacy and Safety of HIP2101 in Patients With Acute or Chronic Gastritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-ESOL-301
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Gastritis
MeSH Terms: conditions — Gastritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIP2101 (Experimental): Taking HIP2101+HPP2102 once daily for 2 weeks.
  Interventions: Drug: HIP2101; Drug: HPP2102
- RLD2101 (Active Comparator): Taking RLD21012101+HPP2101 once daily for 2 weeks.
  Interventions: Drug: RLD2101; Drug: HPP2101

INTERVENTIONS:
Drug: HIP2101 — Test drug
  Arms: HIP2101
Drug: RLD2101 — Reference drug
  Arms: RLD2101
Drug: HPP2101 — Placebo drug
  Arms: RLD2101
Drug: HPP2102 — Placebo drug
  Arms: HIP2101

SUMMARY:
The purpose of this study is to investigate the safety and clinical efficacy of HIP2101 in patients with acute or chronic gastritis.

ELIGIBILITY:
Inclusion Criteria:

* 19≤ age ≤ 75
* Have been diagnosed as acute or chronic gastritis with at least 1 erosion by endoscopy within 7 days before enrollment.
* Patients understood the consents and purpose of this trial and signed consent form

Exclusion Criteria:

* Patients who cannot perform endoscopy
* Active gastric or duodenal ulcer
* Reflux esophagitis, barrett's esophagus, gastric or esophageal varix
* Zollinger-Ellison syndrome, pyloric obstruction, and esophageal stricture, Inflammatory Bowel Diease, acute pancreatitis
* History of gastrointestinal surgery
* History of malignancy tumor, especially in the upper gastrointestinal tract
* Severe liver disorder(at screening day, AST or ALT level exceeds 3 times more than normal upper range)
* Severe renal disorder(at screening day, MDRD eGFP ≤ 30 mL/min/1.73m2) or chronic renal disease
* Bleeding disorder
* Patients who have taken drugs containing following list within 2 weeks before endoscopy : H2-receptor antagonists, Proton pump inhibitors, P-CABs, gastrin inhibitors, antacids, gastric mucosal protectants, anticholinergics
* Patients who have taken anticoagulants within a week before endoscopy
* Patients who have taken drugs containing following list after endoscopy : GI tract regulators, salicylates, steroids, , NSAIDs, bisphosphonates, selective serotonin reuptake inhibitors, iron supplements, oriental herbal medicines
* History of allergic reaction to the medications used in this study
* Use of other investigational drugs within 30 days prior to the study
* History of alcohol or drug abuse
* Positive to pregnancy test, nursing mother, intention on pregnancy
* Considered by investigator as not appropriate to participate in the clinical study with other reason

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Improvement rate of erosion | week 2
  percentage of subjects whose erosion score is improved by more than 50%

SECONDARY OUTCOMES:
Cure rate of erosion | week 2
  percentage of subjects whose erosion is completely cured
Cure rate of edema | week 2
  percentage of subjects whose edema is completely cured
Improvement rate of erythema | week 2
  percentage of subjects whose erythema score is improved by more than 50%
Improvement rate of hemorrage | week 2
  percentage of subjects whose hemorrage score is improved by more than 50%
Improvement rate of GI symptoms | week 2
  percentage of subjects whose GI symptoms score is improved by more than 50%

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim H, Lee JY, Kwon YH, Moon HS, Park JK, Kim KB, Kim SW, Youn YH, Kim SG, Kim GH, Kim JW, Jang JY, Kwon KS, Kwon JG, Kim HS, Hong SJ, Lee KJ, Choi SC, Moon JS, Kim N, Park JJ, Lim Y, Hong SH, Jung HY. Evaluation of the Efficacy and Safety of a Dual Delayed-Release Formulation of 10-mg Esomeprazole in Patients with Gastric Erosions: A Multicenter, Randomized, Double-Blind, Active-Control, Phase III Study. Gut Liver. 2025 Jul 15;19(4):519-527. doi: 10.5009/gnl240390. Epub 2025 Feb 14. PMID 39949051